CLINICAL TRIAL: NCT03915054
Title: Effect of the CAPA Culture Step on Meiotic and Developmental Competence of Human Oocytes After Using Two (Previously Used) Meiotic Maturation Triggers in a SIBLING Oocyte Study Design
Brief Title: Amphiregulin Versus Non-Amphiregulin Supplementation to Maturation Culturing Medium in IVM.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS/BVMD/19/03
Record Dates: First submitted 2019-04-03; First posted 2019-04-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: PCOS; IVM

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AREG-TRIGGER (Active Comparator): Per case (6mL) 5940 µL "Basal Medium"
  * 60 µL "IVM MIX" Do not need to filtrate media.
  Interventions: Drug: AREG-TRIGGER
- CONTROL-TRIGGER (Active Comparator): Per case (5 mL) 4.3 ml IVM Medicult Medium (Vial 2) 0.5 ml HSA (from stock 10% solution) 50µl FSH (from stock 7.5 IU/ml) 5µl hCG (from stock 100 IU/ml) 75 µl GH (from stock 0.66mg/ml)
  Interventions: Drug: CONTROL-TRIGGER

INTERVENTIONS:
Drug: AREG-TRIGGER — Oocytes in AREG-TRIGGER medium will be mature in AREG + FSH + HSA + Insulin + Estradiol medium.
  Per case (6mL) 5940 µL "Basal Medium"
  * 60 µL "IVM MIX" Do not need to filtrate media.
  Other Names: Capacitation IVM medium
  Arms: AREG-TRIGGER
Drug: CONTROL-TRIGGER — Oocytes in CONTROL-TRIGGER medium will be mature in FSH + hCG + GH + HSA medium.
  Per case (5 mL) 4.3 ml IVM Medicult Medium (Vial 2) 0.5 ml HSA (from stock 10% solution) 50µl FSH (from stock 7.5 IU/ml) 5µl hCG (from stock 100 IU/ml) 75 µl GH (from stock 0.66mg/ml)
  Other Names: CAPA Control Medium
  Arms: CONTROL-TRIGGER

SUMMARY:
Clinical use of IVM was pioneered in the nineties, but has not yet become a realistic option for wide-scale practice, for several reasons. Fundamentally, despite recent progress in improving the implantation and the pregnancy rates using in-vitro matured oocytes, results of IVM remain lower than treatment cycles utilizing conventional ART. To improve the outcome of IVM cycles, this study focuses on improving in-vitro culture conditions.

In-vitro maturation (IVM) of human oocytes obtained from minimally stimulated or unstimulated ovaries offers a more "patient friendly" treatment option than the conventional Assisted Reproductive Technology (ART) treatment with controlled ovarian hyperstimulation (COH). Typically, IVM will be offered to women with polycystic ovaries (PCO/PCOS), or to patients with an excellent ovarian reserve, i.e. a high antral follicle count. IVM treatment is characterized by minimal administration of FSH or hMG and NO hCG trigger. The IVM approach is less disruptive to patients' daily life through the reduced need for hormonal and ultrasound monitoring, avoids a range of minor and major complications, such as ovarian hyperstimulation syndrome, and aims to reduce the total cost of infertility treatment for the patient and for the health care budget.

Human oocytes retrieved from small antral follicles are able to resume meiosis by undergoing germinal vesicle breakdown and extrusion of the first polar body, if oocytes have reached meiotic competence. These oocytes can be fertilized although only a proportion (less than 50%) of them can develop further into viable embryos. It has been hypothesized that failure of embryonic development may, at least in part, be due to an immature oocyte cytoplasm. A novel human in vitro maturation (IVM) culture system (named CAPACITATION-IVM is being investigated, hereafter named "CAPA") using 1°) natural compounds known to influence cAMP levels within the cumulus-oocyte-complex and 2°) compounds that are crucial for the oocyte-cumulus cross-talk. Keeping cyclic AMP high after retrieval in the GV oocyte prevents the occurrence of nuclear maturation, enabling increased communication between the oocyte and the cumulus cells. This allows for the improvement in the synchronization of nuclear and cytoplasmic maturation processes in the oocyte, to the benefit of embryo quality.

DETAILED DESCRIPTION:
There are two types of patients can be distinguished in this study:

* Polycystic ovarian morphology + normal cycle length (up to 35 days). The majority of subjects in this group have non-syndromic polycystic ovaries and do not have PCOS. In these patients, AMH is only moderately elevated and cyclical follicular development occurs under the influence of FSH.
* PCOS - Polycystic ovarian morphology + oligomenorrhoea (menstrual periods occurring at intervals of greater than 35 days, with only four to nine periods in a year) or amenorrhea. In these patients, with often strongly elevated AMH levels and concomitant hyperandrogenemia, relative FSH resistance results in arrest of follicular growth at the small antral follicular state. Spontaneous selection of a dominant follicle does not occur or occurs rarely. A large proportion of follicles are atretic. An important proportion of these patients have a BMI higher than 25. These patients generally receive the same standard gonadotropin stimulation regimen as the patients of the previous group, but if the largest follicles have a diameter of less than 8 mm on the third day of stimulation, patients receive one or two supplementary days of gonadotropin stimulation. Moreover, these patients generally take two-three weeks of OCP before the start of the IVM cycle and start stimulation approximately on day five after OCP withdrawal. However, since these patients do not have endogenous FSH-driven recruitment of follicles, the start of stimulation is rather flexible.
* The use of OCP (oral contraceptive pill) before the IVM cycle is obligate. OCP (for example Microgynon 30 micrograms) will be administered daily, to clear the atretic follicles in the ovary. OCP will be given for between 14 and 21 days (this method allows for better programming the cycles and the workload in the embryology lab).

Before the first IVM cycle (Screening visit): All subjects will undergo a pelvic ultrasound scan to evaluate suitability to undergo IVM treatment. Patients will undergo a blood test for serology (Hepatitis B, HIV, syphilis) and baseline hormonal profiling (LH, FSH, E2, progesterone, AMH, SHBG, Testosterone). Additional analysis of TSH, thyroperoxidase antibodies, prolactin. Any concomitant medication taken in the last 3 months prior to the IVM attempt should be notified.

First IVM treatment cycle:

* First clinic visit:

  * All subjects will contact the study nurse on cycle day (cd1) to initiate the first Capacitation culture cycle. If cd1 is during the weekend, subjects will contact the study nurse on Monday. The subject will attend the clinic on day 1, 2 or 3 of menstrual bleeding. An ultrasound scan is performed to rule out the existence of ovarian cysts and a blood sample is taken for hormonal assessment (HCG, FSH, LH, E2, progesterone). On the evening of cycle day 3 of the first clinic visit, flexible Gonadotrophin stimulation will be started to enhance follicular development. The first dose of HP-hMG 150 IU at 2 PM. Second dose next day of HP-hMG 150 IU at 2 PM. The subject will return for a pelvic ultrasound scan and a blood test (FSH, LH, E2, progesterone) after the two days of HP-hMG 150 IU stimulation (i.e. on the morning of day 6).
  * To patients with OCP bleeding: On day one, two, three, or four of the withdrawal bleeding that occurs after discontinuing the OCP, the subject will attend the clinic to undergo a pelvic ultrasound scan and a blood sample is taken for hormonal assessment (FSH, LH, E2, progesterone, AMH, total serum testosterone, SHBG). On the day of the first clinic visit, flexible HP-hMG stimulation will be started to enhance follicular development, at a first daily dose of HP-hMG at 8 P.M. The subject will return for a pelvic ultrasound scan and a blood test (FSH, LH, E2, progesterone) after two days of HP hMG stimulation.
* Second clinic visit at day 6 (after 2 days of HP-hMG treatment):

  * If the ultrasound scan shows the presence of a single dominant follicle larger than 12 mm with the other follicles all less than 10 mm, and the oocyte retrieval (OR) will be scheduled two days later, between 8:00 and 9:00 h. It is important to keep the OR 42 - 46 hours after the last HP-hMG injection as a fixed timing. If the ultrasound scan shows a maximal follicular diameter of less than 8 mm, a final injection of HP-hMG will be administered at 2 P.M. and the oocyte retrieval (OR) will be scheduled two days later, between 8:00 and 9:00 h. It is important to keep the OR 42 - 46 hours after the last HP-hMG injection as a fixed timing.
  * To patients with OCP bleeding: If the ultrasound scan shows a maximal follicular diameter of approx. 9 mm, a final injection of HP-hMG will be administered at 2 P.M. and the oocyte retrieval (OR) will be scheduled two days later, between 8:00 and 9:00 h (under general anesthetics - the exact time of OR should be discussed with operating nurses and anesthetist). It is important to keep the time of OR constant at 42 -46 hours after the last HP-hMG injection.
* Third visit - Oocyte retrieval: Oocyte retrieval (OR) will be scheduled between 8:00 and 10:00 h (under general anesthetics). On the day of OR:

  * An ultrasound scan of both ovaries and of endometrial lining is recorded.
  * A blood sample will be obtained for hormonal profiling (LH, FSH, E2, progesterone).
* All cumulus-oocyte complexes (COC) retrieved from the patient are cultured in CAPA medium for 24 hours.
* Following CAPA culture, half of oocytes will be divided randomly (50/50) to the two maturation triggers medium.

  * Group 1: Medicult IVM media + AREG+FSH+HSA+Insulin+Estradiol (AREG-TRIGGER group)
  * Group 2: Medicult IVM media + FSH+GH+hCG+HSA (CONTROL-TRIGGER group) with no AREG added
* In vitro oocyte maturation:

  * Evaluate and register COCs for cumulus mass (CM) and cumulus contact between oocyte and cumulus cells. Each time take photographs. Discard fully denuded, degenerated oocytes.
  * Transfer half of the COCs (5-10 at a time) from the Capacitation culture dish to the "washing dish" containing "Maturation Medium 1 (AREG-TRIGGER medium)" by using an Eppendorf micropipette and wash them thoroughly (load pipette tips with 5µl, max. 10µl). Then transfer COCs to the "IVM dish" with "Maturation Medium 1 (AREG-TRIGGER medium)".
  * Transfer the second half of the COCs from the Capacitation culture dish to the "washing dish" containing "Maturation Medium 2 (CONTROL-TRIGGER medium)" and wash them thoroughly (load pipette tips with 5µl, max. 10µl). Then transfer COCs to the "IVM dish" with "Maturation Medium 2 (CONTROL-TRIGGER medium)".
  * Keep COCs in pools of ~10.
  * Label the dish appropriately and culture COCs 30-32 hours in an incubator.
* Evaluation of maturation (MII, GVBD, GV) will be done at 30 hours. Oocytes which have undergone GVBD but with no clear PB will be assessed at 32 hours. Insemination will be performed using intra-cytoplasmic sperm injection (3-4 hours after oocyte retrieval or maturation check); only matured oocytes will be inseminated.
* Fertilization check will be performed under an inverted microscope at 16-18 hours after insemination. Embryo evaluation will be performed at 68 ±1 hours after fertilization using the Istanbul consensus. Standard Embryo Vitrification protocol used. Embryos will be vitrified per stimulation protocol obtained (group 1 AREG-TRIGGER or group 2 - CONTROL-TRIGGER).
* Frozen embryo transfer: The patient will be randomized to receive embryo randomly from AREG-TRIGGER or CONTROL-TRIGGER. Where no embryo(s) from the randomized group were available, embryo(s) from the other group were transferred.
* The first pregnancy test was performed 14 days after embryo transfer; a positive pregnancy test was defined as serum beta hCG >5 mIU/mL
* Clinical pregnancy was defined as at least one gestational sac on ultrasound at 7 weeks' gestation with the detection of heartbeat activity.
* Ongoing pregnancy was defined as pregnancy with a detectable heart rate at ≥12 weeks' gestation after the completion of the first transfer.
* Live birth was defined as the birth of at least one newborn after 24 weeks' gestation exhibiting any sign of life (twins were a single count).
* After a first unsuccessful IVM cycle: The clinical and embryological data and results related to the first IVM cycle (cumulative fresh and frozen embryo cycles) will be discussed, to establish a more patient-tailored approach for an eventual second IVM cycle. The patient-tailored approach in the second IVM cycle might consist of modification of the management of the follicular phase.

ELIGIBILITY:
Inclusion Criteria:

* Having polycystic ovarian morphology: at least 24 follicles in both ovaries and/or increased ovarian volume (>10ml) (it is sufficient that 1 ovary fits these criteria)
* Undergoing ≤ 2 previous IVM or IVF attempts
* Agreeing to have ≤ 2 embryos transferred

Exclusion Criteria:

* High grade endometriosis
* Oocyte donation and pre-implantation genetic diagnosis cycles
* Cases with extremely poor sperm quality.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Meiotic maturation efficiency | Two days after oocytes pick-up
  Percentage of PB, GVBD, GV by the two types of trigger. The PB (or MII) oocyte displays the first PB in the PVS. GVBD oocytes have neither a visible GV nor PBI. GV oocyte presents an intracytoplasmic nucleus called the 'germinal vesicle'.
Number of transferable day 3 embryos | Five days after oocytes pick-up
  Number of transferable day 3 embryos obtained by the two meiotic trigger types

SECONDARY OUTCOMES:
Ongoing pregnancy rate | At a minimum of 12 weeks from the beginning of the last menstrual cycle (each cycle is 4 weeks) up to the time of delivery
  Pregnancy with detectable heart rate at 12 weeks' gestation up to the time of delivery
Live birth rate | At least 24 weeks of gestation up to the time of delivery
  Live birth is defined as the birth of at least one newborn after 24 weeks' gestation that exhibits any sign of life (twin will be a single count). For the timing of this occur, ongoing pregnancy will be used, i.e. ongoing pregnancy at 12 weeks will be used in calculations, conditional on the fact that this ongoing pregnancy results in live birth.
Genetic and epigenetic analysis of cord blood of newborns (Will be done in a separate study) | 1 day (Prior to the initiation of IVF/IVM) and 1 day (at the time of delivery)
  Newborn's material (cord blood) will be collected for genetics (karyotyping) and epigenetics analysis.
Genetic and epigenetic analysis of cells from buccal smears of newborns (Will be done in a separate study) | 1 day (Prior to the initiation of IVF/IVM) and 1 day (at the time of delivery)
  Newborn's material (cells from buccal smears) will be collected for genetics (karyotyping) and epigenetics analysis.
Genetic and epigenetic analysis of placenta of newborns (Will be done in a separate study) | 1 day (Prior to the initiation of IVF/IVM) and 1 day (at the time of delivery)
  Newborn's material (placenta) will be collected for genetics (karyotyping) and epigenetics analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD,MCE, Principal Investigator — Hope Research Center
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akin N, Le AH, Ha UDT, Romero S, Sanchez F, Pham TD, Nguyen MHN, Anckaert E, Ho TM, Smitz J, Vuong LN. Positive effects of amphiregulin on human oocyte maturation and its molecular drivers in patients with polycystic ovary syndrome. Hum Reprod. 2021 Dec 27;37(1):30-43. doi: 10.1093/humrep/deab237. PMID 34741172